CLINICAL TRIAL: NCT05311878
Title: Non-invasive Brain Computer Interface for Cognitive Enhancement
Brief Title: Non-invasive BCI for Cognitive Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jose del R. Millan, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020030073_p2
Record Dates: First submitted 2022-02-22; First posted 2022-04-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects; Neuropsychiatric Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EEG based perceptual training (Experimental): Subjects complete a perceptual learning task in which EEG-based visual feedback is provided
  Interventions: Device: EEG-based perceptual training
- Behavior based perceptual training (Active Comparator): Subjects complete a perceptual learning task in which ground truth visual feedback is provided
  Interventions: Device: Behavior based perceptual training

INTERVENTIONS:
Device: EEG-based perceptual training — Electroencephalography (EEG) signals will be recorded from subjects as they perform rotation-based perceptual tasks. The neural correlates of conscious perception of rotations will be processed and decoded in real-time using machine learning algorithms to provide feedback. Subjects are instructed to assume a mental state/find a strategy to maximise the accuracy of feedback. In total, each subject will complete 5 sessions of perceptual training with this intervention.
  Arms: EEG based perceptual training
Device: Behavior based perceptual training — Subjects complete the rotation-based perceptual tasks, and ground truth visual feedback is provided indicating whether subjects have spotted the rotations correctly. Subjects are instructed to spot as many rotation as possible to maximise the accuracy of feedback. In total, each subject will complete 5 sessions of perceptual training with this intervention.
  Arms: Behavior based perceptual training

SUMMARY:
People's perceptual skills can significantly affect their abilities to make optimal decisions, judgments, and actions in real-world dynamic environments. Perceptual learning refers to training and experiences to induce improvements in the ability to make sense of what people see, hear, feel, taste or smell based on ambiguous sensory information. In this study, investigators hypothesise that there exist neural signatures that robustly encode the conscious visual perception of rotations of a cursor and the magnitudes of these rotations in a novel, rotation-based perceptual learning task. Investigators also hypothesise that online, instantaneous EEG-based feedback on subjects' visual perceptions of rotations with an EEG-based Brain Computer Interface (BCI) can foster perceptual learning much more effectively than behaviour perceptual training, especially in very small rotation magnitudes that represent extremely difficult perceptual tasks.

ELIGIBILITY:
Inclusion Criteria:

Able-bodied volunteers:

* good general health
* normal or corrected vision
* no history of neurological/psychiatric disease
* ability to read and understand English
* ability to understand information and ability to give a free and informed consent

Subjects with neuropsychiatric diseases

* Subjects with neuropsychiatric diseases such as bipolar disorder and schizophrenia.
* normal or corrected vision
* ability to read and understand English
* ability to understand information and ability to give a free and informed consent

Exclusion Criteria:

* short attentional spans or cognitive deficits that prevent to remain concentrated during the experimental sessions
* concomitant serious illnesses (e.g., metabolic disorders, cardiac arrest)
* factors hindering proper EEG acquisition (e.g., scalp wound, uncontrolled muscle activity)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in correct answer rate of different rotation magnitudes across 5 intervention sessions | Difference is measured every 24 hours, before versus after each intervention session
  The correct answer rate per rotation magnitude reflects the improvements in perceptual skills across the two conditions. It measures the percentage of each rotation magnitude spotted correctly. The score is 0-100, and the higher the value, the better the outcome.

SECONDARY OUTCOMES:
Change in neural correlates of conscious perception across 5 intervention sessions | Difference is measured every 24 hours, before versus after each intervention session
  This outcome measures whether neural correlates of conscious perception (e.g. amplitude, peak-to-peak, band power and connectivity measures of neural correlates) change across sessions as a result of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jose del R. Millan, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- Engineering Education and Research Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available by the online publication date. These data will be placed in public servers for any interested researcher to access it